CLINICAL TRIAL: NCT03001011
Title: A Randomized, Double Blind, Parallel Group Study For Assessing The Efficacy And Safety Of Renvela® Tablets For The Treatment Of Hyperphosphatemia In Patients With Chronic Kidney Disease Not On Dialysis Versus Placebo
Brief Title: Evaluation of Renvela in Patients With Chronic Kidney Disease Not On Dialysis And Hyperphosphatemia In China
Acronym: RECOVER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14011; U1111-1161-9850 (Other: UTN)
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo (for Renvela) orally 3 times per day (TID) for up to 8 weeks. One to five tablets were taken with meals, as directed by physician and were titrated (up to a maximum of 15 tablets per day) to reach a target goal of serum phosphorus less than or equal to (<=) 4.6 mg/dL (<=1.49 mmol/L).
  Interventions: Drug: Placebo
- Renvela (Experimental): Participants received Renvela orally TID for up to 8 weeks. One to five tablets were taken with meals, as directed by physician and were titrated (up to a maximum of 15 tablets per day) to reach a target goal of serum phosphorus <=4.6 mg/dL (<=1.49 mmol/L).
  Interventions: Drug: Sevelamer Carbonate (GZ419831)

INTERVENTIONS:
Drug: Placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo
Drug: Sevelamer Carbonate (GZ419831) — Pharmaceutical form: tablet
  Route of administration: oral
  Other Names: Renvela
  Arms: Renvela

SUMMARY:
Primary Objective:

To demonstrate efficacy of Renvela tablets in the reduction of serum phosphorus in hyperphosphatemia in participants with chronic kidney disease not on dialysis.

Secondary Objectives:

To document the efficacy of Renvela tablets in the reduction of serum lipids (total cholesterol and low-density lipoprotein cholesterol [LDL-C]).

To document the efficacy of Renvela tablets in the reduction of calcium-phosphorus product.

To document the efficacy of Renvela tablets in the reduction of intact parathyroid hormone (iPTH).

To document the efficacy of Renvela tablets in proportion of participants reaching the target serum phosphorus level 4.6 milligrams per decilitre (mg/dL) (1.47 millimoles per litre [mmol/L], inclusive).

To evaluate safety of Renvela tablets.

DETAILED DESCRIPTION:
The total duration of study period per participant was up to 14 weeks.

ELIGIBILITY:
Inclusion criteria:

* Participants with chronic kidney disease who had not been on dialysis, and were not expected to begin dialysis, or renal transplantation in the next 4 months from the screening visit.
* Had serum phosphorus measurement greater than or equal to (>=) 5.5 mg/dL (1.78 mmol/L) at screening visit (if participants were not on phosphate binder[s] at Screening Visit) OR at the end of Washout Period (if participants were on phosphate binder[s] at screening visit).
* Had the following laboratory measurements at screening visit:

  * 25-hydroxy vitamin D >=10 nanograms per milliliter (ng/mL).
  * intact parathyroid hormone, intact parathyroid hormone (iPTH) <=800 picograms per millilitre (pg/mL).
  * Signed written informed consent.

Exclusion criteria:

* Men or women below 18 years of age.
* Any technical/administrative reason that made it impossible to randomize the participant in the study.
* Was not of the level of understanding and willingness to cooperate with all visits and procedures, as described in the study protocol.
* Not yet received chronic kidney disease diet education before screening visit.
* Not willing and not able to avoid changes to diet during the study.
* Not willing or able to maintain screening doses of lipid lowering medication, 1, 25 dihydroxy vitamin D, and/or cinacalcet for the duration of the study, except for safety reasons.
* Not willing or not able to avoid antacids and phosphate binders containing aluminium, magnesium, calcium, or lanthanum for the duration of the study unless prescribed as an evening calcium supplement.
* Had participated in any other investigational drug studies within 30 days, or 5 half lives, whichever is longer, prior to screening visit.
* Conditions/situations such as:

  * Participant was the Investigator or any Subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
  * Uncooperative or any condition that could make the participant potentially non-compliant to the study procedures (for example, participants could not be contacted by phones as required in phone call visits).
  * Evidence of active malignancy.
  * Not on stable medical condition (for example, but not limited to, active ethanol or drug abuse [tobacco use acceptable]; documented poorly controlled diabetes mellitus, poorly controlled hypertension, active vasculitis, human immunodeficiency virus [HIV] infection), or had any clinically significant medical conditions.
* Had known hypersensitivity to sevelamer or any constituents of Renvela tablets.
* Had bowel obstruction, active dysphagia or swallowing disorder, or a predisposition to or current bowel obstruction, ileus, or severe gastrointestinal motility disorders including severe constipation.
* Using or plan to use anti-arrhythmic or anti-seizure medications for arrhythmia or seizure disorders.
* Was pregnant or breast-feeding.
* If the participant was female, and of childbearing potential (pre-menopausal and not surgically sterile), was not willing to use an effective contraceptive method throughout the study.
* Had any condition, which in the opinion of the investigator would prohibit the participant's inclusion in the study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (38):
- China (38):
  - Investigational Site Number 1560003, Beijing
  - Investigational Site Number 1560026, Cangzhou
  - Investigational Site Number 1560015, Changchun
  - Investigational Site Number 1560011, Changsha
  - Investigational Site Number 1560030, Chongqing
  - Investigational Site Number 1560019, Dalian
  - Investigational Site Number 1560013, Fuzhou
  - Investigational Site Number 1560001, Guangzhou
  - Investigational Site Number 1560027, Guangzhou
  - Investigational Site Number 1560037, Guilin
  - Investigational Site Number 1560031, Haikou
  - Investigational Site Number 1560036, Hengyang
  - Investigational Site Number 1560039, Hengyang
  - Investigational Site Number 1560023, Hohhot
  - Investigational Site Number 1560033, Kunming
  - Investigational Site Number 1560034, Kunming
  - Investigational Site Number 1560006, Lanzhou
  - Investigational Site Number 1560004, Nanchang
  - Investigational Site Number 1560005, Nanchang
  - Investigational Site Number 1560032, Nanchang
  - Investigational Site Number 1560017, Nanjing
  - Investigational Site Number 1560029, Nanning
  - Investigational Site Number 1560028, Ningbo
  - Investigational Site Number 1560002, Shanghai
  - Investigational Site Number 1560007, Shanghai
  - Investigational Site Number 1560021, Shenyang
  - Investigational Site Number 1560038, Shenyang
  - Investigational Site Number 1560025, Shijiazhuang
  - Investigational Site Number 1560022, Taiyuan
  - Investigational Site Number 1560012, Tianjin
  - Investigational Site Number 1560014, Tianjin
  - Investigational Site Number 1560010, Wuhan
  - Investigational Site Number 1560008, Xi'an
  - Investigational Site Number 1560020, Xiamen
  - Investigational Site Number 1560018, Xiamen
  - Investigational Site Number 1560035, Xuzhou
  - Investigational Site Number 1560024, Yinchuan
  - Investigational Site Number 1560016, Zhanjiang

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 38 centers in China. A total of 482 participants were screened between 07 June 2017 & 30 May 2019, of which 280 participants were screen failures. Screen failures were mainly due to serum phosphorus level greater than or equal to >=5.5 milligrams per deciliter (mg/dL) (1.78 millimoles per litre [mmol/L]) at screening visit.
Pre-assignment Details: A total of 202 participants were randomized in the study. Randomization was stratified according to screening serum phosphorus level (>=5.5 - 6.0 mg/dL [1.78 - 1.94 mmol/L] and >6.0 mg/dL [1.94 mmol/L]). Assignment to arms was done centrally using interactive voice/web response system in 1:1 ratio (Renvela [sevelamer carbonate]: placebo).
Period: Overall Study
Arm/Group | Placebo | Renvela
Started | 101 | 101
Completed | 74 | 80
Not Completed | 27 | 21
Not completed — Adverse Event | 9 | 3
Not completed — Chronic kidney disease lead to dialysis | 15 | 10
Not completed — Other than specified above | 3 | 8

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized participants.
Groups:
- Placebo: Participants received placebo (for Renvela) orally TID for up to 8 weeks. One to five tablets were taken with meals, as directed by physician and were titrated (up to a maximum of 15 tablets per day) to reach a target goal of serum phosphorus <= 4.6 mg/dL (<=1.49 mmol/L).
- Total: Total of all reporting groups
Arm/Group | Placebo | Renvela | Total
Number analyzed (Participants) | 101 | 101 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (12.4) | 50.6 (13.5) | 50.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 48 | 94
  Male | 55 | 53 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 101 | 101 | 202
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Phosphorus at Week 8
Description: Baseline of serum phosphorus value was the last serum phosphorus level obtained before the first double-blind investigational medicinal product (IMP) dosing. Missing Week 8 data were imputed by last observation carried forward [LOCF] method.
Time Frame: Baseline, Week 8
Population: Modified intention to treat (mITT) population: all participants who were randomized, received at least 1 dose of IMP & had both baseline assessment & at least 1 post-baseline assessment of phosphorus measure. Here, number analyzed = participants with available data at specified time points.
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 93 | 98
mmol/L
  Baseline | 2.090 [1.870 to 2.270] | 2.095 [1.870 to 2.400]
  Change at Week 8: number analyzed (Participants) | 91 | 97
  Change at Week 8 | 0.010 [-0.200 to 0.250] | -0.200 [-0.490 to 0.020]
Statistical Analysis 1: Comparison: Placebo vs Renvela; A hierarchical testing procedure was used to control type I error & handle multiple secondary endpoint analyses. Testing was then performed sequentially in order outcome measures (OM) are reported. The hierarchical testing sequence continued only when previous OM was statistically significant at 0.05 level; Test type: Superiority; p < 0.0001, Wilcoxon rank sum test — Threshold for statistical significance at 0.05; Median difference (Renvela - Placebo) = -0.210 — Renvela Vs. Placebo

2. Secondary Outcome: Change From Baseline in Total Cholesterol at Week 8
Description: Missing Week 8 data were imputed by LOCF method.
Time Frame: Baseline, Week 8
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 82 | 89
mmol/L | -0.115 [-1.82 to 1.54] | -0.830 [-4.45 to 0.74]

3. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 8
Description: Missing Week 8 data were imputed by LOCF method.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 81 | 86
mmol/L | -0.030 [-1.61 to 1.30] | -0.830 [-3.31 to 0.51]

4. Secondary Outcome: Change From Baseline in Calcium-Phosphorus Product at Week 8
Description: Missing Week 8 data were imputed by LOCF method.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Median (Full Range); unit: mmol^2/L^2
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 90 | 97
mmol^2/L^2 | 0.0200 [-2.648 to 2.936] | -0.4960 [-2.592 to 2.696]

5. Secondary Outcome: Change From Baseline in Intact Parathyroid Hormone (Ipth) Level at Week 8
Description: Missing Week 8 data were imputed by LOCF method.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Median (Full Range); unit: nanogram per liter (ng/L)
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 91 | 97
nanogram per liter (ng/L) | 7.2380 [-298.732 to 573.306] | 0.0000 [-370.172 to 327.966]

6. Secondary Outcome: Percentage of Participants Reaching the Target Serum Phosphorus Level (4.6 mg/dL [1.49 mmol/L]) at Week 8
Description: Missing Week 8 data were imputed by LOCF method.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 91 | 97
percentage of participants | 6.6 | 15.5

7. Secondary Outcome: Change From Baseline in Serum Phosphorus Level at Week 4
Description: Missing Week 4 data were imputed by LOCF method.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 91 | 97
mmol/L | -0.020 [-1.56 to 2.42] | -0.240 [-1.03 to 1.39]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an Adverse Event (AE) without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during TEAE period. On-treatment period was defined as the (time from the first dose of IMP to the last dose of IMP+3 days). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: From first dose of IMP to the last dose of IMP +3 days i.e. up to Day 59
Population: Analysis was performed on safety population that consisted of all randomized participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 101 | 101
Participants
  Any TEAE | 86 | 83
  Any Treatment emergent SAE | 31 | 26
  any TEAE leading to permanent discontinuation | 21 | 12

9. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Hematological Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Hemoglobin: <=115 g/L (Male[M]) or <=95 g/L (Female [F]); >=185 g/L (M) or >=165 g/L (F); Decrease from baseline (DFB) >=20 g/L
  * Hematocrit: <=0.37 v/v (M) or <=0.32 v/v (F); >=0.55 v/v (M) or >=0.5 v/v (F)
  * Red blood cells (RBC): >=6 Tera/L
  * Platelets: <100 Giga/L; >=700 Giga/L
  * White blood cells (WBC): <3.0 Giga/L (Non-Black [NB]) or <2.0 Giga/L (Black [B]); >=16.0 Giga/L
  * Neutrophils: <1.5 Giga/L (NB) or <1.0 Giga/L (B); <1.0 Giga/L
  * Lymphocytes: >4.0 Giga/L
  * Monocytes: >0.7 Giga/L
  * Basophils: >0.1 Giga/L
  * Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN >=0.5 Giga/L)
Time Frame: From first dose of IMP to the last dose of IMP +3 days i.e. up to Day 59
Population: Analysis was performed on safety population. Here, number analyzed = participants with available data for the specified categories.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received placebo (for Renvela) orally TID for up to 8 weeks. One to five tablets were taken with meals, as directed by physician and were titrated (up to a maximum of 15 tablets per day) to reach a target goal of serum phosphorus <= 4.6 mg/dL [<=1.49 mmol/L]).
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 101 | 101
Participants
  Hemoglobin <=115 g/L (M) or <=95 g/L (F): number analyzed (Participants) | 78 | 84
  Hemoglobin <=115 g/L (M) or <=95 g/L (F) | 59 | 54
  Hemoglobin >=185 g/L (M) or >=165 g/L (F): number analyzed (Participants) | 78 | 84
  Hemoglobin >=185 g/L (M) or >=165 g/L (F) | 0 | 0
  Hemoglobin DFB >=20 g/L: number analyzed (Participants) | 78 | 84
  Hemoglobin DFB >=20 g/L | 9 | 6
  Hematocrit <=0.37 v/v (M) or <=0.32 v/v (F): number analyzed (Participants) | 77 | 82
  Hematocrit <=0.37 v/v (M) or <=0.32 v/v (F) | 68 | 67
  Hematocrit >0.55 v/v (M) or >=0.5 v/v (F): number analyzed (Participants) | 77 | 82
  Hematocrit >0.55 v/v (M) or >=0.5 v/v (F) | 0 | 0
  RBC >=6 Tera/L: number analyzed (Participants) | 77 | 83
  RBC >=6 Tera/L | 0 | 1
  Platelets <100 Giga/L: number analyzed (Participants) | 76 | 83
  Platelets <100 Giga/L | 3 | 4
  Platelets >=700 Giga/L: number analyzed (Participants) | 76 | 83
  Platelets >=700 Giga/L | 0 | 0
  WBC <3.0 Giga/L (NB) or <2.0 Giga/L (B): number analyzed (Participants) | 76 | 84
  WBC <3.0 Giga/L (NB) or <2.0 Giga/L (B) | 2 | 0
  WBC >=16.0 Giga/L: number analyzed (Participants) | 76 | 84
  WBC >=16.0 Giga/L | 0 | 0
  Neutrophils <1.5 Giga/L (NB) or <1.0 Giga/L (B): number analyzed (Participants) | 76 | 82
  Neutrophils <1.5 Giga/L (NB) or <1.0 Giga/L (B) | 0 | 0
  Lymphocytes >4 Giga/L: number analyzed (Participants) | 76 | 82
  Lymphocytes >4 Giga/L | 0 | 0
  Monocytes >0.7 Giga/L: number analyzed (Participants) | 76 | 82
  Monocytes >0.7 Giga/L | 0 | 0
  Basophils >0.1 Giga/L: number analyzed (Participants) | 75 | 82
  Basophils >0.1 Giga/L | 0 | 0
  Eosinophils >0.5 Giga/L or >ULN (ULN >=0.5 Giga/L): number analyzed (Participants) | 75 | 82
  Eosinophils >0.5 Giga/L or >ULN (ULN >=0.5 Giga/L) | 4 | 6

10. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Metabolic Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Glucose: <=3.9 mmol/L and < lower limits of normal (LLN); >=11.1 mmol/L (unfasted [unfas]) or >=7 mmol/L (fasted [fas])
  * Triglycerides: >=4.6 mmol/L
  * Albumin: <= 25 g/L.
Time Frame: From first dose of IMP to the last dose of IMP +3 days i.e. up to Day 59
Population: Analysis was performed on safety population. Here, number analyzed = participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 101 | 101
Participants
  Triglycerides: >=4.6 mmol/L: number analyzed (Participants) | 78 | 84
  Triglycerides: >=4.6 mmol/L | 0 | 2
  Glucose: =< 3.9 mmol/L and < LLN: number analyzed (Participants) | 77 | 86
  Glucose: =< 3.9 mmol/L and < LLN | 1 | 1
  Glucose: >=11.1 mmol/L(unfas); >=7 mmol/L(fas): number analyzed (Participants) | 77 | 86
  Glucose: >=11.1 mmol/L(unfas); >=7 mmol/L(fas) | 5 | 6
  Albumin: <= 25 g/L: number analyzed (Participants) | 91 | 97
  Albumin: <= 25 g/L | 1 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Electrolytes
Description: Criteria for potentially clinically significant abnormalities:
  Sodium: <=129 millimoles (mmol)/L; >=160 mmol/L Potassium: <3 mmol/L; >=5.5 mmol/L Chloride: <80 mmol/L; >115 mmol/L.
Time Frame: From first dose of IMP to the last dose of IMP +3 days i.e. up to Day 59
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 101 | 101
Participants
  Sodium <=129 mmol/L: number analyzed (Participants) | 80 | 86
  Sodium <=129 mmol/L | 1 | 3
  Sodium >=160 mmol/L: number analyzed (Participants) | 80 | 86
  Sodium >=160 mmol/L | 0 | 0
  Potassium <3 mmol/L: number analyzed (Participants) | 85 | 93
  Potassium <3 mmol/L | 0 | 0
  Potassium >=5.5 mmol/L: number analyzed (Participants) | 85 | 93
  Potassium >=5.5 mmol/L | 36 | 46
  Chloride <80 mmol/L: number analyzed (Participants) | 92 | 97
  Chloride <80 mmol/L | 0 | 2
  Chloride >115 mmol/L: number analyzed (Participants) | 92 | 97
  Chloride >115 mmol/L | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Renal Function Parameters
Description: Criteria for potentially clinically significant abnormalities:
  Creatinine: >=150 micromol/L; >=30% change from baseline, >=100% change from baseline Creatinine clearance: <15 mL/min; >=15 to <30 mL/min; >=30 to <60 mL/min; >=60 to <90 mL/min Blood urea nitrogen: >=17 mmol/L Uric acid: <120 micromol/L; >408 micromol/L Glomular Filtration Rate (GFR): < 15 mL/min/1.73m^2, >= 15 - < 30 mL/min/1.73m^2, >= 30 - < 60 mL/min/1.73m^2, >= 60 - < 90 mL/min/1.73m^2.
Time Frame: From first dose of IMP to the last dose of IMP +3 days i.e. up to Day 59
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 101 | 101
Participants
  Creatinine >=150 micromol/L: number analyzed (Participants) | 84 | 89
  Creatinine >=150 micromol/L | 84 | 89
  Creatinine >=30% change from baseline: number analyzed (Participants) | 84 | 89
  Creatinine >=30% change from baseline | 15 | 33
  Creatinine >=100% change from baseline: number analyzed (Participants) | 84 | 89
  Creatinine >=100% change from baseline | 3 | 3
  Creatinine Clearance <15 mL/min: number analyzed (Participants) | 84 | 89
  Creatinine Clearance <15 mL/min | 77 | 81
  Creatinine clearance >=15 to <30 mL/min: number analyzed (Participants) | 84 | 89
  Creatinine clearance >=15 to <30 mL/min | 6 | 8
  Creatinine clearance >=30 to <60 mL/min: number analyzed (Participants) | 84 | 89
  Creatinine clearance >=30 to <60 mL/min | 1 | 0
  Creatinine clearance >=60 to <90 mL/min: number analyzed (Participants) | 84 | 89
  Creatinine clearance >=60 to <90 mL/min | 0 | 0
  Blood Urea Nitrogen >=17 mmol/L: number analyzed (Participants) | 79 | 85
  Blood Urea Nitrogen >=17 mmol/L | 77 | 83
  Uric acid <120 micromol/L: number analyzed (Participants) | 80 | 86
  Uric acid <120 micromol/L | 0 | 0
  Uric acid >408 micromol/L: number analyzed (Participants) | 80 | 86
  Uric acid >408 micromol/L | 56 | 67
  GFR < 15 mL/min/1.73m^2: number analyzed (Participants) | 84 | 89
  GFR < 15 mL/min/1.73m^2 | 82 | 86
  GFR >= 15 - < 30 mL/min/1.73m^2: number analyzed (Participants) | 84 | 89
  GFR >= 15 - < 30 mL/min/1.73m^2 | 2 | 3
  GFR >= 30 - < 60 mL/min/1.73m^2: number analyzed (Participants) | 84 | 89
  GFR >= 30 - < 60 mL/min/1.73m^2 | 0 | 0
  GFR >= 60 - < 90 mL/min/1.73m^2: number analyzed (Participants) | 84 | 89
  GFR >= 60 - < 90 mL/min/1.73m^2 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Liver Function Parameters
Description: Criteria for potentially clinically significant abnormalities:
  Alanine Aminotransferase (ALT): >3 ULN; >5 ULN; >10 ULN; Aspartate aminotransferase (AST): >3 ULN.
Time Frame: From first dose of IMP to the last dose of IMP +3 days i.e. up to Day 59
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 101 | 101
Participants
  ALT >3 ULN: number analyzed (Participants) | 77 | 85
  ALT >3 ULN | 1 | 0
  ALT >5 ULN: number analyzed (Participants) | 77 | 85
  ALT >5 ULN | 1 | 0
  ALT >10 ULN: number analyzed (Participants) | 77 | 85
  ALT >10 ULN | 0 | 0
  AST >3 ULN: number analyzed (Participants) | 76 | 85
  AST >3 ULN | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Criteria for potentially clinically significant vital sign abnormalities:
  Systolic blood pressure (SBP) supine: <=95 millimeters of mercury (mmHg) and DFB >=20 mmHg; >=160 mmHg and increase from baseline (IFB) >=20 mmHg Diastolic blood pressure (DBP) supine: <=45 mmHg and DFB >=10 mmHg; >=110 mmHg and IFB >=10 mmHg Heart rate (HR) supine: <=50 beats per minute (bpm) and DFB >=20 bpm; >=120 bpm and IFB >=20 bpm Weight: >=5% DFB; >=5% IFB.
Time Frame: From first dose of IMP to the last dose of IMP +3 days i.e. up to Day 59
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Renvela
Number analyzed (Participants) | 101 | 101
Participants
  SBP (supine) <=95 mmHg and DFB >=20 mmHg: number analyzed (Participants) | 92 | 97
  SBP (supine) <=95 mmHg and DFB >=20 mmHg | 0 | 0
  SBP (supine) >=160 mmHg and IFB >=20 mmHg: number analyzed (Participants) | 92 | 97
  SBP (supine) >=160 mmHg and IFB >=20 mmHg | 17 | 12
  DBP (supine) <=45 mmHg and DFB >=10 mmHg: number analyzed (Participants) | 92 | 97
  DBP (supine) <=45 mmHg and DFB >=10 mmHg | 0 | 0
  DBP (supine) >=110 mmHg and IFB >=10 mmHg: number analyzed (Participants) | 92 | 97
  DBP (supine) >=110 mmHg and IFB >=10 mmHg | 2 | 3
  HR (supine) <=50 bpm and DFB >= 20 bpm: number analyzed (Participants) | 92 | 97
  HR (supine) <=50 bpm and DFB >= 20 bpm | 0 | 0
  HR (supine) >=120 bpm and IFB >=20 bpm: number analyzed (Participants) | 92 | 97
  HR (supine) >=120 bpm and IFB >=20 bpm | 0 | 0
  Weight >=5% DFB: number analyzed (Participants) | 92 | 97
  Weight >=5% DFB | 12 | 7
  Weight >=5% IFB: number analyzed (Participants) | 92 | 97
  Weight >=5% IFB | 14 | 9

ADVERSE EVENTS:
Time Frame: Reported AEs are TEAEs that is AEs that developed/worsened or became serious during the TEAE period (time from the first dose of IMP to the last dose of IMP+3 days i.e. Day 59).
Description: Analysis was performed on safety population.
Groups:
- Placebo: Participants received placebo (for Renvela) orally TID with meals up to 8 weeks as directed by physician and were titrated to reach a target goal of serum phosphorus <=4.6 mg/dL (<=1.49 mmol/L).
- Renvela: Participants received Renvela orally TID with meals up to 8 weeks as directed by physician and were titrated to reach a target goal of serum phosphorus <=4.6 mg/dL (<=1.49 mmol/L).
Arm/Group | Placebo | Renvela
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/101
Serious Adverse Events (participants affected / at risk) | 31/101 | 26/101
Other Adverse Events (participants affected / at risk) | 52/101 | 60/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Renvela (N=101)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2) | 2 (2)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myofascitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 4 (4) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 13 (14) | 8 (8)
Diabetic Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
End Stage Renal Disease (Renal and urinary disorders) | 7 (8) | 9 (9)
Glomerulonephritis Chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arteriovenous Fistula Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Renvela (N=101)
Abdominal Distension (Gastrointestinal disorders) | 5 (5) | 6 (7)
Constipation (Gastrointestinal disorders) | 5 (5) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 5 (5)
Nausea (Gastrointestinal disorders) | 15 (15) | 10 (11)
Vomiting (Gastrointestinal disorders) | 13 (17) | 12 (20)
Oedema Peripheral (General disorders) | 9 (10) | 14 (14)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (9) | 8 (8)
Decreased Appetite (Metabolism and nutrition disorders) | 11 (13) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 18 (24) | 25 (31)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (8) | 3 (3)
Metabolic Acidosis (Metabolism and nutrition disorders) | 7 (7) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT03001011/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT03001011/SAP_001.pdf